CLINICAL TRIAL: NCT01617590
Title: A 48-week, Multi-center, Randomized, Open-lable, Controlled Study to Assess the Response (ACR20) Using Different Disease-Modifying Antirheumatic Drugs Cycle Combination Regimen in Adult Patients With Active Rheumatoid Arthritis
Brief Title: Disease-Modifying Antirheumatic Drugs Cycle Combination Therapy Research
Acronym: DCCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanxi Medical University (Other)
Responsible Party: Principal Investigator, Li Xiaofeng, dean, Shanxi Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DMARD-RA
Record Dates: First submitted 2012-05-28; First posted 2012-06-12 (Estimated); Last update posted 2012-06-14 (Estimated); Status verified 2012-06

CONDITIONS: Rheumatoid Arthritis
Keywords: RA; Leflunomide; Methotrexate
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Leflunomide; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- leflunomide (Experimental): Leflunomide 10-20 mg/d
  Interventions: Drug: leflunomide
- methotrexate (Active Comparator): MTX 7.5-15 mg/week
  Interventions: Drug: methotrexate

INTERVENTIONS:
Drug: leflunomide — Leflunomide 10-20 mg, orally, once daily for up to 48 weeks. Twelve weeks after the initial Leflunomide induction, patients were randomized into two groups (LEF+CTX:LEF+MTX=2:1) if the DAS 28 were higher than 2.6, or continuing leflunomide use without dosing change. Then, the disease activity was assessed using DAS 28 every 12 weeks. The regimen should remain unchanged if the DAS 28 reached to less than 2.6, otherwise, a third (24 weeks) or fourth (36 weeks) DMARs should be added.
  Intravenous CTX was administrated once 200-400mg per 3 weeks.
  Arms: leflunomide
Drug: methotrexate — MTX 7.5-15 mg, orally, once weekly for up to 48 weeks. Twelve weeks after the initial MTX induction, patients were randomized into two groups (MTX+CTX:LEF+MTX=2:1) if the DAS 28 were higher than 2.6, or continuing MTX use without dosing change. Then, the disease activity was assessed using DAS 28 every 12 weeks. The regimen should remain unchanged if the DAS 28 reached to less than 2.6, otherwise, a third (24 weeks) or fourth (36 weeks) DMARs should be added.
  Intravenous CTX was administrated once
  Arms: methotrexate

SUMMARY:
This study was intended to assess the efficacy and safety of different Disease-Modifying Antirheumatic Drugs cycle combination regimen using the American College of Rheumatology (ACR) criteria of 20% improvement in symptoms (ACR20) in managing active adult rheumatoid arthritis.

ELIGIBILITY:
Inclusion Criteria:

RA patients：

* Male and female patients aged 18 - 75 years (inclusive).
* Body weight between 50 and 100 kg (inclusive).
* Post menopausal or surgically sterile female patients are allowed. Female patients of child-bearing potential may participate if they are already on a stable dose of methotrexate. Additional birth control details to be provided at screening. Male patients must use an effective contraception method during the study and at least for 2 months following the completion/discontinuation of the study.
* Diagnosis of RA, classified by American Rheumatism Association 1987 revised criteria.
* Active disease evaluation (DAS 28 > 3.2).
* Patients who using steroids before enrollment, the dose should not be more than 30mg/d, and remain unchanged for more than 30days.
* Without use of other disease activity controlling drugs.
* Get the informed consent.

Exclusion Criteria:

* Advanced patients with severe joints disability.
* Pregnant or breast- feeding female patients.
* Patients with severe primary disease or impairment of heart, brain, lung, liver (ALT or AST > 1.5 normal value), kidney (sCr > normal value), endocrine, and hematology system.
* Concomitant with other rheumatic disease.
* Alcohol taken or drug abusing patients.
* Patients with congestive heart failure, QT prolongation syndrome or poorly controlled diabetes mellitus. Patients with a history of QTc prolongation will be excluded.
* Patients who have received intra-articular or systemic corticosteroid injections having been required for treatment of acute RA flare (not being part of a regular therapeutic regimen) within 4 weeks prior to randomization.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2012-05; Primary Completion 2013-12 (Estimated); Study Completion 2014-05 (Estimated)

PRIMARY OUTCOMES:
ACR20 | 48 weeks
  Percentage of subjects who meet the response rate of ACR20 at each post-dose visit

SECONDARY OUTCOMES:
ACR50 | 48 weeks
  Percentage of subjects who meet the response rate of ACR 50 at week 48
ACR70 | 48week
  Percentage of subjects who meet the response rate of ACR 70 at week 48
EULAR response：good response | 48 week
  Percentage of subjects who meet the EULAR response criteria of good response at week 48
EULAR response ：moderate response | 48 week
  Percentage of subjects who meet the EULAR response criteria of moderate response at week 48

CONTACTS AND LOCATIONS:
Overall Officials: li xiao feng, Principal Investigator — Second Hospital of Shanxi Medical University
Locations (1):
- rheumatism department,Second hospital of Shanxi medical university, Taiyuan, Shanxi, China